CLINICAL TRIAL: NCT04349995
Title: Amplatzer PFO Occluder Post-marketing Surveillance Study
Acronym: PFO PMS Jpn
Status: Active, not recruiting | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: ABT-CIP-10278
Record Dates: First submitted 2020-04-14; First posted 2020-04-16 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: PFO - Patent Foramen Ovale
MeSH Terms: conditions — Foramen Ovale, Patent

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Amplatzer PFO Occluder: Percutaneous PFO Closure using Amplatzer PFO occluder
  Interventions: Device: Amplatzer PFO Occluder

INTERVENTIONS:
Device: Amplatzer PFO Occluder — Percutaneous PFO closure using Amplatzer PFO Occluder

SUMMARY:
The purpose of the Amplatzer PFO Occluder post-marketing clinical use surveillance study is to observe the frequency, type and degree of adverse device effects and adverse events in order to assure the safety of the new medical device, and to collect safety and efficacy information for evaluating the results of the clinical use.

DETAILED DESCRIPTION:
Based on the Ministerial Ordinance on Good Post-marketing Study Practice for Medical Device, the Surveillance will register patients with patent foramen ovale (PFO) who have experienced a PFO-related cryptogenic cerebral infarction (including diagnosed paradoxical cerebral embolism) or transient ischemic attack (determined by positive head imaging such as DWI) in whom an Amplatzer PFO Occluder implant was attempted (Marketing Approval No. 30100BZX00024000, date May 28, 2019, hereinafter referred to as "PFO occluder").

ELIGIBILITY:
Inclusion Criteria:

* Refer to Amplatzer PFO occluder IFU

Exclusion Criteria:

* Refer to Amplatzer PFO occluder IFU

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be considered registered upon insertion of the Amplatzer PFO Occluder delivery system into the body
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2026-05-28 (Estimated)

PRIMARY OUTCOMES:
device- or procedure related SAE rate | up to 30 Days
  device- or procedure related serious adverse events (SAEs) through 30 days
PE, DVT and ischemic stroke and atrial fibrillation rate | beyond 30 days through 3 years
  rate of pulmonary embolism (PE), deep vein thrombosis (DVT), ischemic stroke and atrial fibrillation beyond 30 days through 3 years
Effective PFO closure | At 1 year
  Effective closure of the PFO at 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Abbott Medical Japan LLC, Mita, Minato, Japan

IPD SHARING:
Plan to Share IPD: Undecided